CLINICAL TRIAL: NCT06227156
Title: A Multicenter Open Phase II to Evaluate the Safety, Efficacy and Pharmacokinetic Characteristics of Disitamab Vedotin in the Treatment With HER2- Expression, Subjects With Locally Advanced or Metastatic Castration-resistant Prostate Cancer
Brief Title: Disitamab Vedotin in the Treatment With HER2- Expression, Subjects With Locally Advanced or Metastatic Castration-resistant Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C034
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-01

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: Metastatic Castration-resistant prostate cancer.; HER2- expression
MeSH Terms: interventions — disitamab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin (Experimental): Disitamab Vedotin Q2W arm
  Interventions: Drug: Disitamab Vedotin Injection

INTERVENTIONS:
Drug: Disitamab Vedotin Injection — 2.0 mg/kg, intravenous infusion，D1, every 2 weeks is a treatment cycle
  Other Names: DV,RC48

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Disitamab Vedotin in the treatment of subjects with locally advanced or metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This is a Multicenter Open Phase II to Evaluate the Safety, Efficacy and Pharmacokinetic Characteristics of Disitamab Vedotin in the Treatment With HER2- Expression, Subjects with locally advanced or metastatic castration-resistant prostate cancer.

The study plans to enroll 40 subjects with locally advanced or metastatic CRPC with HER2 expression (IHC 1+ and above) who have been treated with androgen deprivation therapy and novel hormone therapy. Eligible subjects were enrolled and received RC48 intravenous infusion at a dose of 2.0 mg/kg every 2 weeks. Subjects received medication until disease progression, intolerable toxicity, active withdrawal, death, or study termination by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Pathology confirmed prostate adenocarcinoma
3. Locally advanced or metastatic prostate cancer
4. PCWG3 criteria-compliant prostate cancer progression occurs during androgen deprivation therapy (or bilateral scrotal excision). Progression will be determined based on at least 1 of the following criteria: PSA progression: defined as 2 consecutive increases in PSA, separated by at least 1 week, relative to the previous reference value. If a confirmed PSA increase is the only indicator of progression, then 1 ng/mL is the minimum starting value; Soft tissue progression: defined as an increase of ≥20% in the sum of the diameters of all target lesions (short-axis for lymph node lesions and long-axis for non-lymph node lesions) relative to the sum of the smallest diameters at the start of treatment or the presence of one or more new lesions; Bone lesion progression: defined as the detection of at least two additional new lesions on bone scan.
5. Serum testosterone level ≤ 50 ng/dL (or ≤ 1.73 nmol/L), prior to the first study drug administration;
6. Continuous androgen deprivation therapy (ADT) with LHRH agonists or LHRH antagonists or previous bilateral orchiectomy (surgical debridement) during the study period;
7. Confirmed HER2 expression (IHC 1+, 2+, 3+), HER2 gene amplification, or HER2 gene mutation;
8. Subjects were able to provide paraffin blocks or at least 5 paraffin embedded sections (white pieces) for HER2 detection, and the presence of HER2 expression was confirmed by central laboratory tests (immunohistochemistry 1+, 2+, 3+)；
9. Previous medical androgen deprivation therapy (or bilateral scrotal excision) and new hormone therapy (e.g. abiraterone, enzalutamide) and have developed disease progression
10. The following criteria should be met within 7 days prior to the first study dose:

    1. haemoglobin ≥ 9 g/dL;
    2. absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
    3. platelet count ≥ 100 × 109/L;
    4. serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN);
    5. without liver metastasis, alanine aminotransferase and aspartate aminotransferase ≤ 2.5 × ULN; with liver metastasis, alanine aminotransferase and aspartate aminotransferase ≤ 5 × ULN;;
    6. albumin (ALB) ≥ 25 g/L;
    7. blood creatinine ≤ 1.5 × ULN, or calculated according to the Cockcroft-Gault formula, creatinine clearance (CrCl) ≥ 50 mL/min;
    8. left ventricular ejection fraction (LVEF) ≥ 50%;
11. ECOG Physical Status Score of 0-1
12. Expected survival ≥ 6 months
13. Subjects whose spouses are of childbearing age must agree to use contraception during the study and for 6 months after the last dose; sperm donation is not permitted during the study and for 6 months after the last dose
14. Ability to understand and sign an informed consent form.

Exclusion Criteria:

1. Systematic chemotherapy, novel hormone therapy, targeted therapy, immunotherapy, or other antitumor therapy (including 5-alpha reductase inhibitors, oestrogens, and medroxyprogesterone, etc.)was administered prior to the initial study drug, and treatment ended within 5 half-lives (or 2 weeks, whichever is shorter) of the initial study drug. Except maintenance castration therapy (LHRH agonists or LHRH antagonists) or bone metastasis therapy(e.g., denosumab, zoledronic acid); In the first study, Chinese medicines with anti-tumor indications were used 2 weeks before administration.
2. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis (subjects who have been treated for brain metastases may be enrolled in this study provided they have stable disease [no evidence of progression as determined by imaging for at least 4 weeks prior to study dosing and and all neurological symptoms have fully recovered], there is no evidence of new or enlarging brain metastases, and discontinuation of steroid therapy at least 7 days prior to the first dose of the trial treatment. (This exception does not include carcinomatous meningitis, which should be excluded regardless of whether it is clinically stable or not).
3. Has received anti-HER2 therapy ;
4. Major surgery, systemic radiotherapy or biologic therapy within 4 weeks prior to first study drug administration, or minor surgery or local radiotherapy within 1 week prior to enrollment;
5. Toxicity due to prior antineoplastic therapy that has not recovered to Common Terminology Criteria for Adverse Events (CTCAE Version 5.0) Grade 1 or below, with the exception of alopecia and abnormalities in laboratory tests or toxicity associated with LHRH agonists or LHRH antagonists that are not considered by the investigator to pose a safety risk;
6. Known allergic reactions to components of the study treatment or its analogues
7. Diagnosis of other malignancies that are expected to affect life expectancy or may interfere with disease assessment. Except for cured non-melanoma skin cancer and superficial bladder cancer
8. Severe and/or persistent infection within 14 days prior to starting the study drug
9. Serum virological tests: positive HBsAg test result with a positive HBV DNA copy number; positive HCVAb test result; positive HIVAb test result;
10. Known serious cardiovascular disease, including any of the following: myocardial infarction, thrombotic event, or unstable angina pectoris in the past 3 months; chronic heart failure, New York Heart Association (NYHA) class II or higher; presence of unstable arrhythmia; uncontrolled hypertension;
11. Combined grade 2 and higher (CTCAE version 5.0) peripheral neuropathy
12. Presence of other systemic diseases that, in the judgement of the investigator, are not under stable control, including diabetes mellitus, liver cirrhosis, pneumonitis, and obstructive pulmonary disease;
13. In the judgement of the investigator, there were other circumstances that made participation in the study unsuitable.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression free survival，rPFS | Up to approximately 2 years
  Define imaging disease progression according to RECIST v1.1 (for all lesions except bone lesions) or PCWG3 (for bone lesions) as the time from the first dose of the drug to the time when the imaging shows disease progression or death.

SECONDARY OUTCOMES:
Objective remission rate (ORR) | Up to approximately 2 years
  ORR assessed according to the evaluation criteria for the efficacy of solid tumors (RECIST 1.1)
Disease Control Rate (DCR) | Until progression, assessed up to approximately 2 years
  Percentage of patients with complete response, partial response, or stable disease for a certain period of time according to RECIST v1.1.
Time to PSA progression(TTPP) | Until progression, assessed up to approximately 2 years
  Defined as time from date of first dose to first PSA progression
Duration of response (DoR) | Until progression, assessed up to approximately 2 years
  Defined as the time from the date of first documented response (CR/PR) until the first progression or death in the absence of disease progression by Investigators assessment according to RECIST 1.1
PSA response rate | Until progression, assessed up to approximately 2 years
  Percent of subjects with different degree of decrease in PSA compared to baseline
Time to first symptomatic bone-related event (SSE) | Until progression, assessed up to approximately 2 years
  Defined as the time from the first dose to the first occurrence of SSE.
Overall Survival (OS) | Up to approximately 2 years
  OS was defined as the time from the date of randomization to the date of death from any cause.
Cmax of RC48 | Up to approximately 2 years
  Peak Plasma Concentration of RC48
AUC of RC48 | Up to approximately 2 years
  Area under the plasma concentration versus time curve of RC48
AUC of MMAE | Up to approximately 2 years
  Area under the plasma concentration versus time curve of MMAE
Immunogenicity of RC48 | up to approximately 2 years
  Anti-drug antibody (ADA) of RC48 positive samples, etc.
Percentage of Participants With Adverse Events (AEs) | Up to approximately 2 years
  Number of participants with adverse effects of treatment. Frequency and severity of adverse effects of treatment as assessed by NCI CTCAE v5.0
Incidence of laboratory tests abnormalities | Up to follow-up period, approximately 2 years
  To be summarized using descriptive statistics
Incidence of ECG abnormalities | Up to follow-up period, approximately 2 years
  To be summarized using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Fang, Ph.D, Study Director — RemeGen Co., Ltd.
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Third Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No